CLINICAL TRIAL: NCT07018193
Title: The Study of Personalized Health Check-up Programs and Standards for High-altitude Migrant Populations
Status: Not yet recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Other Study IDs: PHC-high
Record Dates: First submitted 2025-05-12; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: High Altitude
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exploration group: 200 participants, to explore and formulate and optimize personalized plans and standards for health examinations for people living in plateaus.
- Verification group: 100 participants, to verify the feasibility of the physical examination plan and its effectiveness in the early diagnosis of altitude sickness and plateau environment-related comorbidities.

SUMMARY:
By using wearable devices to monitor and record the physiological data changes and health outcomes (incidence and severity of high-altitude illnesses) of high-altitude migrants at different stages (pre-entry, acute/chronic high-altitude phases, and de-acclimatization phase), and referencing previous cohort studies on high-altitude populations, the study aims to provide a basis for developing personalized health assessment protocols for high-altitude migrants. The formulated assessment protocols and standards will then be validated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥18;
* Those living in plains and preparing to move to the plateau for a short-term or medium-term period;
* Can understand the research requirements and be willing to sign a written informed consent form (ICF).

Exclusion Criteria:

* Past history of contraindicated plateau travel: such as advanced COPD (FEV₁<30% of the expected value or requires continuous oxygen therapy), advanced cystic fibrosis (FEV₁<30% of the expected value or requires continuous oxygen therapy), advanced restricted pulmonary disease (FEV₁<50% of the expected value or requires continuous oxygen therapy), decompensated heart failure, high-risk pregnancy, myocardial infarction or stroke occurred within 90 days, poorly controlled epilepsy, pulmonary hypertension (PASP>90mmHg), sickle cell anemia, unstable angina pectoris, high-risk cerebrovascular abnormalities that have not been treated, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruit those who live in plains and prepare to move to the plateau in the short term or medium term.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of high altitude sickness and related diseases. | through study completion, an average of 3 years
  Early diagnosis rates of acute and chronic altitude sickness and related diseases induced or aggravated by the plateau population in migrant plateau populations.